CLINICAL TRIAL: NCT01106092
Title: Immunogenicity and Reactogenicity of a Booster Dose of GlaxoSmithKline Biologicals' GSK2036874A Vaccine in Healthy Toddlers
Brief Title: Study to Evaluate the Immunogenicity and Reactogenicity of a Booster Dose of GSK2036874A Vaccine in Healthy Toddlers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 113264; 2016-000645-31 (EudraCT Number)
Record Dates: First submitted 2010-04-01; First posted 2010-04-19 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Haemophilus Influenzae Type b; Tetanus; Hepatitis B; Whole Cell Pertussis; Diphtheria; Poliomyelitis Vaccines
MeSH Terms: conditions — Haemophilus Infections; Tetanus; Hepatitis B; Diphtheria

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- GSK2036874A GROUP 1 (Experimental): Healthy male or female children between and including 12 and 24 months of age at the time of the booster vaccination, who were primed with a three-dose vaccination course of polio vaccine, additionally received 1 dose of GSK2036874A vaccine (Formulation 1) intramuscularly into the anterolateral region of the left thigh, at Day 0.
  Interventions: Biological: GSK2036874A vaccine
- GSK2036874A GROUP 2 (Experimental): Healthy male or female children between and including 12 and 24 months of age at the time of the booster vaccination, who were primed with a three-dose vaccination course of polio vaccine, additionally received 1 dose of GSK2036874A vaccine (Formulation 2) intramuscularly into the anterolateral region of the left thigh, at Day 0.
  Interventions: Biological: GSK2036874A vaccine
- GSK2036874A GROUP 3 (Experimental): Healthy male or female children between and including 12 and 24 months of age at the time of the booster vaccination, who were primed with a three-dose vaccination course of polio vaccine, additionally received 1 dose of GSK2036874A vaccine (Formulation 3) intramuscularly into the anterolateral region of the left thigh, at Day 0.
  Interventions: Biological: GSK2036874A vaccine
- ZILBRIX/HIB/POLIORIX GROUP (Active Comparator): Healthy male or female children between and including 12 and 24 months of age at the time of the booster vaccination, who were primed with a three-dose vaccination course of polio vaccine, additionally received 1 dose of Zilbrix/Hib™ and Poliorix™ vaccines at Day 0, administered intramuscularly into the anterolateral regions of the left and right thighs, respectively.
  Interventions: Biological: Zilbrix™/Hib vaccine; Biological: Poliorix™

INTERVENTIONS:
Biological: GSK2036874A vaccine — Intramuscular, single dose
  Arms: GSK2036874A GROUP 1; GSK2036874A GROUP 2; GSK2036874A GROUP 3
Biological: Zilbrix™/Hib vaccine — Intramuscular, single dose
  Arms: ZILBRIX/HIB/POLIORIX GROUP
Biological: Poliorix™ — Intramuscular, single dose
  Arms: ZILBRIX/HIB/POLIORIX GROUP

SUMMARY:
The purpose of the study is to assess the immunogenicity and safety of three formulations of GSK Biologicals' GSK2036874A vaccine compared to Zilbrix™/Hib and Poliorix™ vaccines administered concomitantly, when administered as a single booster dose to healthy poliovirus-primed toddlers aged 12-24 months.

DETAILED DESCRIPTION:
The study will be conducted in a partially double-blinded manner. The study will be double-blinded with respect to the three GSK2036874A formulation groups and open-label with respect to the Control Group.

ELIGIBILITY:
Inclusion Criteria:

* A male or female subject, between and including 12 and 24 months of age at the time of booster vaccination.
* Subjects who have received three doses of polio vaccine as primary vaccination along with the routine vaccinations indicated during the first year of life.
* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative (s) can and will comply with the requirements of the protocol.
* Written informed consent obtained from the parent(s)/Legally Acceptable Representative (s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the booster dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the booster dose.
* Administration of a vaccine not foreseen by the study protocol within 30 days prior to booster vaccination, or planned administration during the active study period (up to Visit 2).
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* History of diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis and/or Haemophilus influenza type b diseases.
* Previous booster vaccination against diphtheria, tetanus, pertussis, poliomyelitis, hepatitis B or H. influenzae diseases.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* A family history of congenital or hereditary immunodeficiency.
* Major congenital defects or serious chronic illness.
* History of neurologic disorders or seizures.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* Administration of immunoglobulins and/or any blood products within the three months preceding the booster dose or planned administration during the study period.
* Occurrence of transient thrombocytopenia or neurological complications following an earlier immunisation against diphtheria and/or tetanus.
* Child in care.
* Occurrence of any of the following adverse events after a previous administration of a diphtheria-tetanus-pertussis vaccine:

  * encephalopathy of unknown aetiology occurring within seven days following previous vaccination with pertussis-containing vaccine,
  * fever >= 40 °C within 48 hours of vaccination not due to another identifiable cause,
  * collapse or shock-like state within 48 hours of vaccination,
  * convulsions with or without fever, occurring within 3 days of vaccination.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature >= 37.5°C on oral, axillary or tympanic setting, or >= 38.0°C on rectal setting.
  * Subjects with a minor illness without fever may, be enrolled at the discretion of the investigator.
* Other conditions which, in the opinion of the investigator, may potentially interfere with interpretation of study results.

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 312 (Actual)
Dates: Start 2010-05-13 (Actual); Primary Completion 2010-09-02 (Actual); Study Completion 2010-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, City of Muntinlupa, Philippines

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Quiambao B, Van Der Meeren O, Kolhe D, Gatchalian S. A randomized, dose-ranging assessment of the immunogenicity and safety of a booster dose of a combined diphtheria-tetanus-whole cell pertussis-hepatitis B-inactivated poliovirus-Hemophilus influenzae type b (DTPw-HBV-IPV/Hib) vaccine vs. co-administration of DTPw-HBV/Hib and IPV vaccines in 12 to 24 months old Filipino toddlers. Hum Vaccin Immunother. 2012 Mar;8(3):347-54. doi: 10.4161/hv.18630. Epub 2012 Feb 14. PMID 22330958
- [Background] Quiambao B et al. The immunogenicity and safety of a new combined DTPw-HBV-IPV/HIB vaccine when administered as a booster dose in Filipino toddlers. Abstract presented at the 7th World Congress for World Society for Pediatric Infectious Diseases (WSPID), Melbourne, Australia, 16-19 November 2011.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 113264 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113264 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113264 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113264 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113264 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113264 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113264 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Period: Overall Study
Arm/Group | GSK2036874A Group 1 | GSK2036874A Group 2 | GSK2036874A Group 3 | Zilbrix/Hib/Poliorix Group
Started | 78 | 78 | 78 | 78
Completed | 78 | 78 | 78 | 77
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2036874A Group 1 | GSK2036874A Group 2 | GSK2036874A Group 3 | Zilbrix/Hib/Poliorix Group | Total
Number analyzed (Participants) | 78 | 78 | 78 | 78 | 312
Age, Continuous [Mean (Standard Deviation); unit: Months] | 17.4 (3.81) | 18 (2.96) | 17.7 (3.38) | 17.5 (3.59) | 17.65 (3.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 31 | 35 | 40 | 143
  Male | 41 | 47 | 43 | 38 | 169
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian-South East Asian heritage | 78 | 78 | 78 | 78 | 312

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects Against Poliovirus Types 1, 2 and 3
Description: Seroprotection was defined as anti-polio types 1, 2 and 3 antibody titres ≥ 8 effective dose (ED50), for 50% of vaccinated subjects.
Time Frame: One month after booster vaccination (At Month 1)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2036874A Group 1 | GSK2036874A Group 2 | GSK2036874A Group 3 | Zilbrix/Hib/Poliorix Group
Number analyzed (Participants) | 78 | 78 | 78 | 77
Participants
  Anti-polio 1 | 78 | 77 | 78 | 77
  Anti-polio 2: number analyzed (Participants) | 77 | 78 | 78 | 77
  Anti-polio 2 | 77 | 78 | 78 | 77
  Anti-polio 3 | 77 | 77 | 78 | 77
Statistical Analysis 1: Comparison: GSK2036874A Group 1 vs Zilbrix/Hib/Poliorix Group; To demonstrate the non-inferiority of GSK2036874A vaccine (Formulation 1) compared to Poliorix™ vaccine co-administered with Zilbrix™/Hib vaccine, in terms of seroprotection rates to the three poliovirus types and to demonstrate that the formulation induces at least a two-fold increase in the geometric mean of the individual ratios (post- over pre-booster titres) for anti-polio type 1 antibodies, one month after vaccination; Test type: Non-Inferiority — Criterion for evaluation of Non-inferiority: The upper limit (UL) of the standardized asymptotic 95% confidence interval (CI) on the group [Zilbrix/Hib/Poliorix Group - GSK2036874A Group 1] difference in percentage of seroprotected subjects ≤ 10%. The lower limit of the asymptotic 95% CI on the geometric mean of the individual ratios (post- over pre-booster titres) for anti-poliovirus type 1 is ≥ 2; Difference in seroprotection rate = 0, 95% CI 2-sided [-4.78 to 4.72]
Statistical Analysis 2: Comparison: GSK2036874A Group 2 vs Zilbrix/Hib/Poliorix Group; To demonstrate the non-inferiority of GSK2036874A vaccine (Formulation 2) compared to Poliorix™ vaccine co-administered with Zilbrix/Hib™ vaccine, in terms of seroprotection rates to the three poliovirus types and to demonstrate that the formulation induces at least a two-fold increase in the geometric mean of the individual ratios (post- over pre-booster titres) for anti-polio type 1 antibodies, one month after vaccination; Test type: Non-Inferiority — Criterion for evaluation of Non-inferiority: The UL of the standardized asymptotic 95% CI on the group [Zilbrix/Hib/Poliorix Group - GSK2036874A Group 2] difference in percentage of seroprotected subjects ≤ 10%. The lower limit of the asymptotic 95% CI on the geometric mean of the individual ratios (post- over pre-booster titres) for anti-poliovirus type 1 is ≥ 2; Difference in seroprotection rate = 1.28, 95% CI 2-sided [-3.53 to 6.94]
Statistical Analysis 3: Comparison: GSK2036874A Group 3 vs Zilbrix/Hib/Poliorix Group; To demonstrate the non-inferiority of GSK2036874A vaccine (Formulation 3) compared to Poliorix™ vaccine co-administered with Zilbrix/Hib™ vaccine, in terms of seroprotection rates to the three poliovirus types and to demonstrate that the formulation induces at least a two-fold increase in the geometric mean of the individual ratios (post- over pre-booster titres) for anti-polio type 1 antibodies, one month after vaccination; Test type: Non-Inferiority — Criterion for evaluation of Non-inferiority: The UL of the standardized asymptotic 95% CI on the group [Zilbrix/Hib/Poliorix Group - GSK2036874A Group 3] difference in percentage of seroprotected subjects ≤ 10%. The lower limit of the asymptotic 95% CI on the geometric mean of the individual ratios (post- over pre-booster titres) for anti-poliovirus type 1 is ≥ 2; Difference in seroprotection rate = 0, 95% CI 2-sided [-4.78 to 4.72]
Statistical Analysis 4: Comparison: GSK2036874A Group 1 vs Zilbrix/Hib/Poliorix Group; To demonstrate the non-inferiority of GSK2036874A vaccine (Formulation 1) compared to Poliorix™ vaccine co-administered with Zilbrix/Hib™ vaccine, in terms of seroprotection rates to the three poliovirus types and to demonstrate that the formulation induces at least a two-fold increase in the geometric mean of the individual ratios (post- over pre-booster titres) for anti-polio type 2 antibodies, one month after vaccination; Test type: Non-Inferiority — Criterion for evaluation of Non-inferiority: The UL of the standardized asymptotic 95% CI on the group [Zilbrix/Hib/Poliorix Group - GSK2036874A Group 1] difference in percentage of seroprotected subjects ≤ 10%. The lower limit of the asymptotic 95% CI on the geometric mean of the individual ratios (post- over pre-booster titres) for anti-poliovirus type 2 is ≥ 2; Difference in seroprotection rate = 0, 95% CI 2-sided [-4.78 to 4.78]
Statistical Analysis 5: Comparison: GSK2036874A Group 2 vs Zilbrix/Hib/Poliorix Group; To demonstrate the non-inferiority of GSK2036874A vaccine (Formulation 2) compared to Poliorix™ vaccine co-administered with Zilbrix/Hib™ vaccine, in terms of seroprotection rates to the three poliovirus types and to demonstrate that the formulation induces at least a two-fold increase in the geometric mean of the individual ratios (post- over pre-booster titres) for anti-polio type 2 antibodies, one month after vaccination; Test type: Non-Inferiority — Criterion for evaluation of Non-inferiority: The UL of the standardized asymptotic 95% CI on the group [Zilbrix/Hib/Poliorix Group - GSK2036874A Group 2] difference in percentage of seroprotected subjects ≤ 10%. The lower limit of the asymptotic 95% CI on the geometric mean of the individual ratios (post- over pre-booster titres) for anti-poliovirus type 2 is ≥ 2; Difference in seroprotection rate = 0, 95% CI 2-sided [-4.78 to 4.72]
Statistical Analysis 6: Comparison: GSK2036874A Group 3 vs Zilbrix/Hib/Poliorix Group; To demonstrate the non-inferiority of GSK2036874A vaccine (Formulation 3) compared to Poliorix™ vaccine co-administered with Zilbrix/Hib™ vaccine, in terms of seroprotection rates to the three poliovirus types and to demonstrate that the formulation induces at least a two-fold increase in the geometric mean of the individual ratios (post- over pre-booster titres) for anti-polio type 2 antibodies, one month after vaccination; Test type: Non-Inferiority — Criterion for evaluation of Non-inferiority: The UL of the standardized asymptotic 95% CI on the group [Zilbrix/Hib/Poliorix Group - GSK2036874A Group 3] difference in percentage of seroprotected subjects ≤ 10%. The lower limit of the asymptotic 95% CI on the geometric mean of the individual ratios (post- over pre-booster titres) for anti-poliovirus type 2 is ≥ 2; Difference in seroprotection rate = 0, 95% CI 2-sided [-4.78 to 4.72]
Statistical Analysis 7: Comparison: GSK2036874A Group 1 vs Zilbrix/Hib/Poliorix Group; To demonstrate the non-inferiority of GSK2036874A vaccine (Formulation 1) compared to Poliorix™ vaccine co-administered with Zilbrix/Hib™ vaccine, in terms of seroprotection rates to the three poliovirus types and to demonstrate that the formulation induces at least a two-fold increase in the geometric mean of the individual ratios (post- over pre-booster titres) for anti-polio type 3 antibodies, one month after vaccination; Test type: Non-Inferiority — Criterion for evaluation of Non-inferiority: The UL of the standardized asymptotic 95% CI on the group [Zilbrix/Hib/Poliorix Group - GSK2036874A Group 1] difference in percentage of seroprotected subjects ≤ 10%. The lower limit of the asymptotic 95% CI on the geometric mean of the individual ratios (post- over pre-booster titres) for anti-poliovirus type 3 is ≥ 2; Difference in seroprotection rate = 1.28, 95% CI 2-sided [-3.53 to 6.94]
Statistical Analysis 8: Comparison: GSK2036874A Group 2 vs Zilbrix/Hib/Poliorix Group; To demonstrate the non-inferiority of GSK2036874A vaccine (Formulation 2) compared to Poliorix™ vaccine co-administered with Zilbrix/Hib™ vaccine, in terms of seroprotection rates to the three poliovirus types and to demonstrate that the formulation induces at least a two-fold increase in the geometric mean of the individual ratios (post- over pre-booster titres) for anti-polio type 3 antibodies, one month after vaccination; Test type: Non-Inferiority — Criterion for evaluation of Non-inferiority: The UL of the standardized asymptotic 95% CI on the group [Zilbrix/Hib/Poliorix Group - GSK2036874A Group 2] difference in percentage of seroprotected subjects ≤ 10%. The lower limit of the asymptotic 95% CI on the geometric mean of the individual ratios (post- over pre-booster titres) for anti-poliovirus type 3 is ≥ 2; Difference in seroprotection rate = 1.28, 95% CI 2-sided [-3.53 to 6.94]
Statistical Analysis 9: Comparison: GSK2036874A Group 3 vs Zilbrix/Hib/Poliorix Group; To demonstrate the non-inferiority of GSK2036874A vaccine (Formulation 3) compared to Poliorix™ vaccine co-administered with Zilbrix/Hib™ vaccine, in terms of seroprotection rates to the three poliovirus types and to demonstrate that the formulation induces at least a two-fold increase in the geometric mean of the individual ratios (post- over pre-booster titres) for anti-polio type 3 antibodies, one month after vaccination; Test type: Non-Inferiority — Criterion for evaluation of Non-inferiority: The UL of the standardized asymptotic 95% CI on the group [Zilbrix/Hib/Poliorix Group - GSK2036874A Group 3] difference in percentage of seroprotected subjects ≤ 10%. The lower limit of the asymptotic 95% CI on the geometric mean of the individual ratios (post- over pre-booster titres) for anti-poliovirus type 3 is ≥ 2; Difference in seroprotection rate = 0, 95% CI 2-sided [-4.78 to 4.72]

2. Primary Outcome: Anti-polio Types 1, 2 and 3 Antibody Titers
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: Prior to booster vaccination (At Month 0)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2036874A Group 1 | GSK2036874A Group 2 | GSK2036874A Group 3 | Zilbrix/Hib/Poliorix Group
Number analyzed (Participants) | 78 | 78 | 78 | 77
Titers
  Anti-polio 1 | 321.1 [231.2 to 446.0] | 219.1 [144.0 to 333.6] | 296.6 [205.1 to 428.8] | 296.9 [213.9 to 412.1]
  Anti-polio 2: number analyzed (Participants) | 77 | 78 | 78 | 77
  Anti-polio 2 | 186.8 [140.1 to 249.2] | 152.2 [111.8 to 207.3] | 183.4 [146.4 to 229.7] | 148.0 [112.4 to 194.9]
  Anti-polio 3 | 74.5 [56.0 to 99.0] | 82.1 [62.1 to 108.6] | 102.1 [77.6 to 134.4] | 79.1 [57.9 to 108.1]

3. Primary Outcome: Anti-polio Types 1, 2 and 3 Antibody Titers
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: One month after booster vaccination (At Month 1)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2036874A Group 1 | GSK2036874A Group 2 | GSK2036874A Group 3 | Zilbrix/Hib/Poliorix Group
Number analyzed (Participants) | 78 | 78 | 78 | 77
Titers
  Anti-polio 1 | 2218.4 [1786.3 to 2755.1] | 1486.7 [1065.9 to 2073.5] | 1245.1 [1007.2 to 1539.2] | 3760.2 [2973.7 to 4754.7]
  Anti-polio 2: number analyzed (Participants) | 77 | 78 | 78 | 77
  Anti-polio 2 | 1598.8 [1293.5 to 1976.3] | 1056.4 [841.5 to 1326.1] | 966.5 [779.5 to 1198.3] | 2883.2 [2275.2 to 3653.8]
  Anti-polio 3 | 2820 [2129.9 to 3733.9] | 2217.7 [1654 to 2973.4] | 1915.8 [1498.1 to 2449.8] | 3626.4 [2618.2 to 5022.9]

4. Secondary Outcome: Number of Seroconverted Subjects for Anti-polio Types 1, 2 and 3
Description: Seroconversion was defined as: For initially seronegative subjects, antibody titer ≥ 8 ED50 one month after the booster dose. For initially seropositive subjects: antibody titer one month after the booster dose ≥ 4 fold the pre-booster antibody titer. For subjects with pre-booster antibody titer below the highest dilution tested (reciprocal < 8192 ED50): highest dilution tested one month after the booster dose (reciprocal > 8192 ED50).
Time Frame: One month after booster vaccination (At Month 1)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2036874A Group 1 | GSK2036874A Group 2 | GSK2036874A Group 3 | Zilbrix/Hib/Poliorix Group
Number analyzed (Participants) | 78 | 78 | 78 | 77
Participants
  Anti-polio 1 | 70 | 64 | 60 | 69
  Anti-polio 2: number analyzed (Participants) | 77 | 78 | 78 | 77
  Anti-polio 2 | 68 | 66 | 70 | 72
  Anti-polio 3 | 74 | 74 | 73 | 75

5. Secondary Outcome: Number of Seroprotected Subjects Against Poliovirus Types 1, 2 and 3
Description: as for outcome 1
Time Frame: Prior to booster vaccination (At Month 0)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2036874A Group 1 | GSK2036874A Group 2 | GSK2036874A Group 3 | Zilbrix/Hib/Poliorix Group
Number analyzed (Participants) | 78 | 78 | 78 | 77
Participants
  Anti-polio 1 | 76 | 70 | 74 | 75
  Anti-polio 2 | 77 | 75 | 78 | 74
  Anti-polio 3 | 74 | 76 | 76 | 70

6. Secondary Outcome: Number of Seroprotected Subjects Against Diphteria (D) and Tetanus (T)
Description: Seroprotection was defined as anti-D and anti-T antibody concentration ≥ 0.1 international units per milliliter (IU/mL).
Time Frame: Prior to (At Month 0) and one month after booster vaccination (At Month 1)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2036874A Group 1 | GSK2036874A Group 2 | GSK2036874A Group 3 | Zilbrix/Hib/Poliorix Group
Number analyzed (Participants) | 78 | 78 | 78 | 77
Participants
  Anti-D, M0 | 69 | 69 | 69 | 65
  Anti-D, M1 | 78 | 78 | 78 | 77
  Anti-T, M0 | 78 | 77 | 77 | 76
  Anti-T, M1 | 78 | 78 | 78 | 77

7. Secondary Outcome: Anti-D and Anti-T Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in IU/mL.
Time Frame: Prior to (At Month 0) and one month after booster vaccination (At Month 1)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | GSK2036874A Group 1 | GSK2036874A Group 2 | GSK2036874A Group 3 | Zilbrix/Hib/Poliorix Group
Number analyzed (Participants) | 78 | 78 | 78 | 77
IU/mL
  Anti-D, M0 | 0.301 [0.237 to 0.382] | 0.331 [0.258 to 0.424] | 0.330 [0.264 to 0.412] | 0.374 [0.276 to 0.508]
  Anti-D, M1 | 6.519 [5.46 to 7.783] | 7.687 [6.112 to 9.669] | 8.659 [7.132 to 10.514] | 6.807 [5.231 to 8.858]
  Anti-T, M0 | 0.776 [0.639 to 0.942] | 0.766 [0.622 to 0.944] | 0.833 [0.668 to 1.038] | 0.932 [0.756 to 1.149]
  Anti-T, M1 | 26.12 [22.65 to 30.121] | 31.047 [25.954 to 37.139] | 31.054 [26.837 to 35.934] | 24.402 [21.042 to 28.298]

8. Secondary Outcome: Number of Seroprotected and Seropositive Subjects for Anti-hepatitis B (Anti-HBs)
Description: Seropositivity was defined as anti-HBs antibody concentration ≥ 3.3 milli-international units per milliliter (mIU/mL). Seprotection was defined as anti-HBs antibody concentration ≥ 10 mIU/mL. Note that percentage of subjects with concentration ≥ 10 mIU/mL was over-estimated due to the use of in-house assay overestimating concentrations between 10-100 mIU/mL. Accordingly GMCs were also overestimated. A decrease in the specificity of the anti-HB ELISA assay had been observed in some studies for low levels of antibody (10-100 mIU/mL). The table shows updated results following partial or complete retesting/reanalysis. Some of the available blood samples initially tested with ELISA were re-tested using the new assay, CLIA.
Time Frame: Prior to (At Month 0) and one month after the booster vaccination (At Month 1)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2036874A Group 1 | GSK2036874A Group 2 | GSK2036874A Group 3 | Zilbrix/Hib/Poliorix Group
Number analyzed (Participants) | 78 | 78 | 78 | 77
Participants
  Anti-HBs ≥ 3.3 mIU/mL, M0 | 71 | 70 | 73 | 73
  Anti-HBs ≥ 3.3 mIU/mL, M1 | 78 | 77 | 78 | 77
  Anti-HBs ≥ 10 mIU/mL, M0 | 64 | 67 | 62 | 70
  Anti-HBs ≥ 10 mIU/mL, M1 | 77 | 77 | 78 | 77

9. Secondary Outcome: Anti-HBs Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in mIU/mL.
Time Frame: Prior to (At Month 0) and one month after the booster vaccination (At Month 1)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK2036874A Group 1 | GSK2036874A Group 2 | GSK2036874A Group 3 | Zilbrix/Hib/Poliorix Group
Number analyzed (Participants) | 78 | 78 | 78 | 77
mIU/mL
  Anti-HBs, M0 | 59.9 [40.3 to 89.1] | 46.9 [32.8 to 67.2] | 61.9 [42.2 to 91] | 88.5 [60.7 to 129]
  Anti-HBs, M1 | 2713.4 [1846.9 to 3986.2] | 2395.1 [1630 to 3519.4] | 3992.8 [2747.2 to 5803.1] | 3484.3 [2452.2 to 4950.8]

10. Secondary Outcome: Number of Seroprotected Subjects Against Polyribosil-ribitol-phosphate (PRP)
Description: Seprotection was defined as anti-PRP antibody concentration ≥ 0.15 micrograms per milliliter (μg/mL).
Time Frame: Prior to (At Month 0) and one month after booster vaccination (At Month 1)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subject for whom immunogenicity data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2036874A Group 1 | GSK2036874A Group 2 | GSK2036874A Group 3 | Zilbrix/Hib/Poliorix Group
Number analyzed (Participants) | 78 | 78 | 78 | 77
Participants
  Anti-PRP, M0 | 28 | 27 | 30 | 35
  Anti-PRP, M1 | 77 | 76 | 71 | 76

11. Secondary Outcome: Anti-PRP Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in μg/mL.
Time Frame: Prior to (At Month 0) and one month after booster vaccination (At Month 1)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | GSK2036874A Group 1 | GSK2036874A Group 2 | GSK2036874A Group 3 | Zilbrix/Hib/Poliorix Group
Number analyzed (Participants) | 78 | 78 | 78 | 77
μg/mL
  Anti-PRP, M0 | 0.134 [0.109 to 0.166] | 0.137 [0.11 to 0.172] | 0.152 [0.118 to 0.197] | 0.171 [0.13 to 0.226]
  Anti-PRP, M1 | 2.871 [1.797 to 4.587] | 2.243 [1.52 to 3.31] | 1.575 [1.065 to 2.33] | 3.305 [2.373 to 4.603]

12. Secondary Outcome: Number of Seropositive Subjects for Anti-Bordetella Pertussis (Anti-BPT)
Description: Seropositivity was defined as anti-BPT antibody concentration ≥ 15 enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: Prior to (At Month 0) and one month after the booster vaccination (At Month 1)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2036874A Group 1 | GSK2036874A Group 2 | GSK2036874A Group 3 | Zilbrix/Hib/Poliorix Group
Number analyzed (Participants) | 76 | 78 | 78 | 77
Participants
  Anti-BPT, M0 | 50 | 50 | 51 | 49
  Anti-BPT, M1: number analyzed (Participants) | 76 | 74 | 77 | 75
  Anti-BPT, M1 | 76 | 73 | 77 | 75

13. Secondary Outcome: Anti-BPT Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in EL.U/mL.
Time Frame: Prior to (At Month 0) and one month after booster vaccination (At Month 1)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK2036874A Group 1 | GSK2036874A Group 2 | GSK2036874A Group 3 | Zilbrix/Hib/Poliorix Group
Number analyzed (Participants) | 76 | 78 | 78 | 77
EL.U/mL
  Anti-BPT, M0 | 19.6 [16.4 to 23.6] | 20.1 [16.5 to 24.5] | 18.9 [15.9 to 22.4] | 19.5 [16 to 23.9]
  Anti-BPT, M1: number analyzed (Participants) | 76 | 74 | 77 | 75
  Anti-BPT, M1 | 161.8 [143.6 to 182.3] | 182.9 [158 to 211.9] | 211 [190.1 to 234.2] | 194.7 [170.6 to 222.4]

14. Secondary Outcome: Number of Subjects With a Booster Response for Anti-BPT
Description: Booster response was defined as: For initially seronegative subjects, antibody concentration ≥ 15 EL.U/mL one month after the booster dose. For initially seropositive subjects: antibody concentration one month after the booster dose ≥ 2 fold the pre-booster antibody concentration.
Time Frame: One month after booster vaccination (At Month 1)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2036874A Group 1 | GSK2036874A Group 2 | GSK2036874A Group 3 | Zilbrix/Hib/Poliorix Group
Number analyzed (Participants) | 74 | 74 | 77 | 75
Participants | 72 | 72 | 77 | 72

15. Secondary Outcome: Number of Subjects With Any Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 8-day (Days 0-7) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2036874A Group 1 | GSK2036874A Group 2 | GSK2036874A Group 3 | Zilbrix/Hib/Poliorix Group
Number analyzed (Participants) | 78 | 78 | 78 | 78
Participants
  Any Pain | 67 | 65 | 66 | 68
  Any Redness | 28 | 29 | 35 | 35
  Any Swelling | 33 | 32 | 36 | 35

16. Secondary Outcome: Number of Subjects With Any Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite and fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 8-day (Days 0-7) post-vaccination period
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2036874A Group 1 | GSK2036874A Group 2 | GSK2036874A Group 3 | Zilbrix/Hib/Poliorix Group
Number analyzed (Participants) | 78 | 78 | 78 | 78
Participants
  Any Drowsiness | 43 | 42 | 46 | 41
  Any Irritability | 53 | 60 | 57 | 65
  Any Loss of appetite | 33 | 36 | 36 | 38
  Any Temperature (Axillary) | 59 | 60 | 57 | 63

17. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Day 0-Day 30) post-vaccination period
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2036874A Group 1 | GSK2036874A Group 2 | GSK2036874A Group 3 | Zilbrix/Hib/Poliorix Group
Number analyzed (Participants) | 78 | 78 | 78 | 78
Participants | 30 | 44 | 30 | 40

18. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Month 0 to Month 1)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2036874A Group 1 | GSK2036874A Group 2 | GSK2036874A Group 3 | Zilbrix/Hib/Poliorix Group
Number analyzed (Participants) | 78 | 78 | 78 | 78
Participants | 1 | 3 | 2 | 1

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms: During the 8-day (Days 0-7) follow-up period after vaccination. Unsolicited AE(s): During the 31-day (Days 0-30) follow-up period after vaccination. SAE(s): During the entire study period (from Month 0 to Month 1).
Arm/Group | GSK2036874A Group 1 | GSK2036874A Group 2 | GSK2036874A Group 3 | Zilbrix/Hib/Poliorix Group
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/78 | 0/78 | 0/78
Serious Adverse Events (participants affected / at risk) | 1/78 | 3/78 | 2/78 | 1/78
Other Adverse Events (participants affected / at risk) | 75/78 | 74/78 | 76/78 | 77/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2036874A Group 1 (N=78) | GSK2036874A Group 2 (N=78) | GSK2036874A Group 3 (N=78) | Zilbrix/Hib/Poliorix Group (N=78)
Febrile convulsion (Nervous system disorders) | 0 | 3 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2036874A Group 1 (N=78) | GSK2036874A Group 2 (N=78) | GSK2036874A Group 3 (N=78) | Zilbrix/Hib/Poliorix Group (N=78)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 10 | 9 | 8
Pain (General disorders) | 67 | 65 | 66 | 68
Redness (General disorders) | 28 | 29 | 35 | 35
Swelling (General disorders) | 33 | 32 | 36 | 35
Drowsiness (General disorders) | 43 | 42 | 46 | 41
Fever (General disorders) | 59 | 60 | 57 | 63
Irritability (General disorders) | 53 | 60 | 57 | 65
Loss of appetite (General disorders) | 33 | 36 | 36 | 38
Nasopharyngitis (Infections and infestations) | 3 | 12 | 11 | 13
Upper respiratory tract infection (Infections and infestations) | 9 | 12 | 5 | 9
Conjunctivitis bacterial (Infections and infestations) | 1 | 4 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.